CLINICAL TRIAL: NCT05142488
Title: Study of Immunogenicity Equivalence After a Homologous Third Dose of Covid-19 (Recombinante) Vaccine, 6 Months After the Second Dose, Comparing Intervals of 8 and 12 Weeks Between the First Two Doses.
Brief Title: Study of Immunogenicity Equivalence of a Homologous Third Dose of Covid-19 (Recombinante) Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ASCLIN 009/2021
Record Dates: First submitted 2021-11-30; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Vaccines

STUDY DESIGN:
Masking Description: Only the laboratory technician will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8 week interval (Experimental): Third dose Covid-19 (recombinante) vaccine 6 months after the second dose of a two dose vaccine schedule with a 8 week interval between the first two doses.
  Interventions: Biological: Covid -19 (recombinante) vaccine
- 12 week interval (Active Comparator): Third dose Covid-19 (recombinante) vaccine 6 months after the second dose of a two dose vaccine schedule with a 12 week interval between the first two doses.
  Interventions: Biological: Covid -19 (recombinante) vaccine

INTERVENTIONS:
Biological: Covid -19 (recombinante) vaccine — Third dose of the Covid-19 (recombinante) vaccine, 6 months after the second dose of a two dose Covid-19 (recombinante) homologous vaccine schedule.

SUMMARY:
The purpose of this study is to evaluate the antibody response, safety and reactogenicity of a third dose Covid-19 (recombinante) vaccine, 6 months after a two-dose vaccine schedule using the same vaccine in all doses.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants giving written informed consent will be evaluated for eligibility criteria. At day 0, participants who meet the eligibility requirements will undergo a thorough medical evaluation and a urine pregnancy test (if applicable). Previous vaccination information will be collected with the participant and checked via digital Covid-19 vaccine certification from the Brazilian public health national immunization program system (SI-PNI) ou from Fundação Oswaldo Cruz (Fiocruz) institutional occupational medicine data. According to the data collected, participants will be placed in one of two groups: 8 or 12 weeks interval between the first two vaccine doses in the vaccine schedule. Eligible and consenting participants will have a blood sample collected and receive immediately after a third dose of the Covid-19 (recombinante) vaccine. Participants will be instructed to fill out an adverse events journal for solicited adverse events for 7 days and non-solicited adverse events for 28 days after the third dose. The research team will contact the participant remotely at least once during the first two weeks. The participant will return for a follow-up visit to the research center 28 days after the third dose, to evaluate adverse events, collect a second blood sample and undergo a thorough medical evaluation. The participant will return to the research center to collect blood samples in three more follow-up visits: 3 months, 6 months and 12 months after the third dose.

ELIGIBILITY:
Inclusion Criteria:

* Employee of Fundação Oswaldo Cruz, stationed in Manguinhos campus, in Rio de Janeiro.
* Previous two-dose vaccine schedule with Covid-19 (recombinante) in both doses, with an interval of8 or 12 weeks between doses.
* A 6-month interval (5 to 7 month window) between the second and the third dose of Covid-19 (recombinante) vaccine.
* Availability to participate during the entire study, and ability to follow study protocol strictly.
* Consent to supply personal contact information, such as telephone numbers, address and other information so the research team may contact the participant (For example, in case the participant fails to attend a scheduled visit without previous notice)
* Ability to understand and sign the volunteered and informed consent form, and ability to fill in the adverse events journal at home, according to the evaluation of the principal investigator ou delegated research team members.
* Understanding the impossibility of participating in another clinical trial while participating in this clinical trial.

Exclusion Criteria:

* Receiving another Covid-19 vaccine after inclusion in the study
* Receiving any vaccine 28 days after administration of a third dose of Covid-19 (recombinante) vaccine.
* Refusal to sign the voluntary and informed consent form or refusal to permit collection of blood samples before the third dose of the Covid-19 (recombinante) vaccine.
* Receiving any other vaccine 28 days before the inclusion in the study
* Previous vaccine schedule with other Covid-19 vaccines, in the first and/or second dose.
* Covid-19 disease confirmed by RT-PCR (Real time polymerase chain reaction) up to 28 days before inclusion in the study.
* Covid-19 symptoms up to 10 days before the inclusion in the study.
* Fever (Axillary temperature above 37,8 º C / 100,04 °F) 72 hours before vaccination in the study.
* Contraindications to the Covid-19 (recombinante) vaccine - Fiocruz/AstraZeneca
* Use of immunosuppressive medication, such as systemic corticosteroids or chemotherapy, or immunosuppressive diseases. We will consider as immunosuppressive doses of systemic corticosteroids daily doses of prednisone of 10mg or more, for more than 14 days.
* Incapacitating mental illness
* Any discoveries made by the principal investigator that would enhance the risk of an adverse result following the participation in the study, or that in some other way justifies exclusion from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 662 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
IgG Anti-S response after a third dose of Covid-19 (recombinante) vaccine | 28 days
  Equivalence of antibody IgG Anti-S response in geometric mean titers, measured immediately before and 28 days after a third dose of Covid-19 (recombinante) vaccine, administered 6 months after the second dose of a two-dose homologous Covid-19 (recombinante) vaccine schedule, between participants with an 8 and 12 week interval between the first two doses.

SECONDARY OUTCOMES:
Duration of Immunogenicity after the third dose of Covid-19 (recombinate) vaccine after 3, 6 and 12 months | 15 months
  Antibody IgG Anti-S collected immediately before, 28 days, 3 months, 6 months and 12 months after the third dose of Covid-19 (recombinante) vaccine.
Safety and reactogenicity of a third dose of Covid-19 (recombinate) vaccine | 15 months
  Safety and reactogenicity after a third dose of Covid-19 (recombinate) vaccine, 7 days for solicited adverse events, 28 days for non-solicited adverse events and 12 months for serious adverse events.
Neutralizing antibodies in plaque reduction neutralization test (PRNT) in a smaller sample | 28 days
  Measure neutralizing antibodies in plaque reduction neutralization test (PRNT) in a smaller sample of participants, immediately before and 28 days after the third dose.
IgG Anti-S response after a third dose of Covid-19 (recombinante) vaccine by age groups | 1 month
  Equivalence of antibody IgG Anti-S response in geometric mean titers, measured immediately before and 28 days after a third dose of Covid-19 (recombinante) vaccine, administered 6 months after the second dose of a two-dose homologous Covid-19 (recombinante) vaccine schedule, between participants with an 8 and 12 week interval between the first two doses. Compare results between participants with 40 years or less, 40 to 60 years, or more than 60 years.
Duration of Immunogenicity after the third dose of Covid-19 (recombinate) vaccine after 3, 6 and 12 months by age groups | 15 months
  Antibody IgG Anti-S collected immediately before, 28 days, 3 months, 6 months and 12 months after the third dose of Covid-19 (recombinante) vaccine. Compare results between participants with 40 years or less, 40 to 60 years, or more than 60 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Unidade de Ensaios Clínicos em Imunobiológicos, Rio de Janeiro, Brazil